CLINICAL TRIAL: NCT04351152
Title: A Phase 3 Randomized, Placebo-Controlled Study of Lenzilumab in Hospitalized Patients With Severe and Critical COVID-19 Pneumonia
Brief Title: Phase 3 Study to Evaluate Efficacy and Safety of Lenzilumab in Patients With COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGEN003-06
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Disease 2019 (COVID-19) Pneumonia
Keywords: Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF); GM-CSF monoclonal antibody; Cytokine Release Syndrome (CRS); Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); Lenzilumab; Cytokine Storm
MeSH Terms: conditions — COVID-19; Pneumonia; Cytokine Release Syndrome | interventions — lenzilumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenzilumab Arm (Experimental): Participants will receive IV infusion of lenzilumab upon randomization at a pre-specified dosing interval and continued administration of standard of care
  Interventions: Biological: Lenzilumab; Drug: Standard of Care
- Placebo Arm (Placebo Comparator): Participants will receive IV infusion of preservative-free 0.9% sodium chloride solution upon randomization matched to lenzilumab at same pre-specified dosing interval and continued administration of standard of care
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Biological: Lenzilumab — Administered as an intravenous (IV) infusion
  Other Names: Humaneered® anti-human GM-CSF monoclonal Antibody
  Arms: Lenzilumab Arm
Drug: Standard of Care — Standard of care therapy can include remdesivir and/or dexamethasone per institutional treatment guidelines or written policies

SUMMARY:
The primary objective of this study is to assess whether the use of lenzilumab in addition to current standard of care can alleviate the immune-mediated cytokine release syndrome (CRS) and improve ventilator-free survival in hospitalized subjects with severe or critical COVID-19 pneumonia.

DETAILED DESCRIPTION:
In COVID-19, high levels of granulocyte macrophage-colony stimulating factor (GM-CSF) and inflammatory myeloid cells correlate with disease severity, cytokine storm, and respiratory failure. The mortality rate for hospitalized COVID-19 patients remains unacceptably high, particularly in patients who progress to invasive mechanical ventilation (IMV). This randomized, double-blind, multicenter, placebo-controlled pivotal phase 3 trial will evaluate the impact of lenzilumab (anti-human GM-CSF monoclonal antibody) on ventilator-free survival in hospitalized, hypoxic patients with COVID-19. The study is also designed to evaluate other key endpoints, including ventilator-free days, duration of ICU stay, incidence of IMV, ECMO and/or death, time to death, all-cause mortality and time to recovery.

Approximately 516 patients will be randomized to receive lenzilumab + SOC vs. placebo + SOC in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older who are capable of providing informed consent or have a proxy capable of giving consent for them
* Virologic confirmation of SARS-CoV-2 infection via any FDA authorized diagnostic test for SARS-CoV-2
* Pneumonia diagnosed by Chest X-ray or Computed Tomography revealing infiltrates consistent with pneumonia
* SpO2 ≤ 94% on room air and/or require low-flow supplemental oxygen and/or require high-flow oxygen support or NIPPV
* Hospitalized, not requiring invasive mechanical ventilation during this hospitalization
* Have not participated in other clinical trial for COVID-19 using an immunomodulatory monoclonal antibody or kinase inhibitor (use of remdesivir, corticosteroids, convalescent plasma, hydroxychloroquine or chloroquine is permitted)
* Females of childbearing potential must have a negative serum or urine pregnancy test

Exclusion Criteria:

* Requiring invasive mechanical ventilation or extracorporeal membrane oxygenation prior to randomization
* Confirmed diagnosis of bacterial pneumonia or other active/uncontrolled fungal or viral infections at screening/baseline
* Known active tuberculosis (TB), history of incompletely treated TB or suspected or known extrapulmonary TB
* Currently receiving treatment for hepatitis A, hepatitis B, hepatitis C or HIV infection
* History of pulmonary alveolar proteinosis (PAP)
* Women of childbearing potential who are pregnant or breastfeeding
* Known hypersensitivity to lenzilumab or any of its components
* Use of any FDA authorized anti-IL-6 (e.g., tocilizumab, sarilumab, sitlukimab), anti-IL-1 (e.g., anakinra, canakinumab), kinase inhibitor (e.g., baracitinib, ibrutinib, acalabrutinib), or neutralizing monoclonal antibody (e.g. bamlanivimab or casirivimab/imdevimab) therapy to treat COVID-19 within 8 weeks prior to randomization
* Use of GM-CSF agents (e.g., sargramostim) within prior 2 months of randomization
* Expected survival < 48h in the opinion of the investigator
* Any condition that, in the opinion of the investigator, is likely to interfere with the safety and efficacy of the study treatment or puts the patient at unacceptably high risk from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free Survival | Up to Day 28

SECONDARY OUTCOMES:
Ventilator-free Days | Up to Day 28
Duration of Intensive Care Unit (ICU) Stay | Up to Day 28
Incidence of Invasive Mechanical Ventilation, ECMO and/or Death | Up to Day 28
Time to Death | Up to Day 28
All-cause Mortality | Day 28
Time to Recovery | Up to Day 28
  Time to recovery is defined as the first day on which a subject satisfies one of the following 3 categories from the 8-point ordinal scale (Hospitalized, not requiring supplemental oxygen-no longer requires ongoing medical care; Not hospitalized, limitation on activities and/or requiring home oxygen; Not hospitalized, no limitations on activities).
Incidence of severe acute respiratory distress syndrome (ARDS) | Up to Day 28
Duration of Hospitalization | Up to Day 28
Time to Improvement in 1 or 2 Categories using 8-point Ordinal Scale | Up to Day 28
Number of Subjects Alive and Off Oxygen | Up to Day 60
Percentage of Participants Experiencing Adverse Events | Up to Day 60
  Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Percentage of Participants Experiencing Serious Adverse Events | Up to Day 60
  Using the NCI CTCAE version 5.0
Proportion of Subjects Discharged from Hospital | Up to Day 60
Time to improvement in oxygenation for > 48 hours | Up to Day 28
Incidence of Non-invasive Ventilation (or Use of High-flow Oxygen Device) | Up to Day 28
Time to Clinical Improvement, Defined as NEWS2 < 2 Maintained for 24 Hours | Up to Day 28
  NEWS2 consists of: Physiological Parameters: respiration rate (per minute), SpO2 Scale 1 (%), SpO2 Scale 2 (%), use of air or oxygen, systolic blood pressure (mmHg), pulse (per minute), consciousness and temperature (°C)
Change from Baseline to Day 28 in Clinical status Based on the 8-point Ordinal Scale | Up to Day 28
Duration of Time on Low-flow or High-flow Supplemental Oxygen | Up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Durrant, MD, Study Director — Humanigen, Inc.
Locations (29):
- United States (18):
  - Mayo Clinic, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - University of Southern California (USC) Medical Center, Los Angeles, California
  - USC - Los Angeles County Medical Center, Los Angeles, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Mercy Medical Center, Rockville Centre, New York
  - Atrium Health, Charlotte, North Carolina
  - St. David's Healthcare, Austin, Texas
  - St. David's North Austin Medical Center, Austin, Texas
  - Texas Health, Dallas, Texas
- Brazil (11):
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - CPCLIN - Centro de Pesquisas Clínicas de Natal, Natal, Rio Grande do Norte
  - Hospital São Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Sociedade Literaria e Caritativa Santo Agostinho, Criciúma, Santa Catarina
  - Hospital Dia do Pulmão, Blumenau, São Paulo
  - Hospital Guilherme Alvaro, Santos, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos LTDA-EPP, São Bernardo do Campo, São Paulo
  - Clinica de Alergia Martti Antila S/S LTDA, Sorocaba, São Paulo
  - Escola Paulista de Medicina (UNIFESP), São Paulo
  - Hospital Heliópolis, São Paulo
  - Hospital São Luiz do Jabaquara/IDOR, São Paulo

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Temesgen Z, Kelley CF, Cerasoli F, Kilcoyne A, Chappell D, Durrant C, Ahmed O, Chappell G, Catterson V, Polk C, Badley A, Marconi VC; LIVE-AIR Study Group. C reactive protein utilisation, a biomarker for early COVID-19 treatment, improves lenzilumab efficacy: results from the randomised phase 3 'LIVE-AIR' trial. Thorax. 2023 Jun;78(6):606-616. doi: 10.1136/thoraxjnl-2022-218744. Epub 2022 Jul 6. PMID 35793833
- [Derived] Temesgen Z, Burger CD, Baker J, Polk C, Libertin CR, Kelley CF, Marconi VC, Orenstein R, Catterson VM, Aronstein WS, Durrant C, Chappell D, Ahmed O, Chappell G, Badley AD; LIVE-AIR Study Group. Lenzilumab in hospitalised patients with COVID-19 pneumonia (LIVE-AIR): a phase 3, randomised, placebo-controlled trial. Lancet Respir Med. 2022 Mar;10(3):237-246. doi: 10.1016/S2213-2600(21)00494-X. Epub 2021 Dec 1. PMID 34863332
- [Derived] Temesgen Z, Burger CD, Baker J, Polk C, Libertin C, Kelley C, Marconi VC, Orenstein R, Durrant C, Chappell D, Ahmed O, Chappell G, Badley AD. LENZILUMAB EFFICACY AND SAFETY IN NEWLY HOSPITALIZED COVID-19 SUBJECTS: RESULTS FROM THE LIVE-AIR PHASE 3 RANDOMIZED DOUBLE-BLIND PLACEBO-CONTROLLED TRIAL. medRxiv [Preprint]. 2021 May 5:2021.05.01.21256470. doi: 10.1101/2021.05.01.21256470. PMID 33972949
- [Derived] Aroldi A, Chiarle R, Gambacorti-Passerini C. Clinical Benefit of Lenzilumab in Cases of Coronavirus Disease 2019. Mayo Clin Proc. 2021 Mar;96(3):817. doi: 10.1016/j.mayocp.2020.12.030. Epub 2021 Jan 11. No abstract available. PMID 33673929
- [Derived] Temesgen Z, Assi M, Shweta FNU, Vergidis P, Rizza SA, Bauer PR, Pickering BW, Razonable RR, Libertin CR, Burger CD, Orenstein R, Vargas HE, Palraj R, Dababneh AS, Chappell G, Chappell D, Ahmed O, Sakemura R, Durrant C, Kenderian SS, Badley AD. GM-CSF Neutralization With Lenzilumab in Severe COVID-19 Pneumonia: A Case-Cohort Study. Mayo Clin Proc. 2020 Nov;95(11):2382-2394. doi: 10.1016/j.mayocp.2020.08.038. Epub 2020 Sep 3. PMID 33153629